CLINICAL TRIAL: NCT05080439
Title: Comparative Effects of Two Conservative Treatments in Teres Major in Handball Athletes With Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Responsible Party: Principal Investigator, Sandra Jiménez, PhD Physiotherapist, University of Valladolid
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: University of Valladolid.
Record Dates: First submitted 2021-09-02; First posted 2021-10-15 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Shoulder Pain; Dry Needling; Diacutaneous Fibrolysis; Athletic Injuries
MeSH Terms: conditions — Shoulder Pain; Athletic Injuries | interventions — Dry Needling

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Diacutaneous Fibrolysis (Experimental): Diacutaneous Fibrolysis in the teres major muscle
  Interventions: Other: Diacutaneous Fibrolysis
- Dry needling (Experimental): Dry needling based on fast-in fast-out technique in the teres major muscle
  Interventions: Other: Dry needling

INTERVENTIONS:
Other: Diacutaneous Fibrolysis — Application of diacutaneous fibrolysis in teres major
  Arms: Diacutaneous Fibrolysis
Other: Dry needling — Dry needling based on fast-in fast-out technique in the teresa major muscle
  Arms: Dry needling

SUMMARY:
The aim of the study is to investigate the effects of the dry needling technique and diacutaneous fibrolysis technique in teres major muscles on pain, range of motion, strength extensibility and muscular properties of the soft tissues of the shoulder in athletes with shoulder pain.

ELIGIBILITY:
Inclusion Criteria:

* Athletes with Shoulder pain
* Glenohumeral internal rotation deficit
* Presence of active MTrP in the teres major muscle

Exclusion Criteria:

* Previous surgery in the upper limb
* Previous physiotherapy treatments in the shoulder
* Dry needling contraindications
* Previous dry needling experience to mantain the blinding

Ages: 18 Years to 35 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2021-09-10 (Actual); Primary Completion 2021-10-31 (Actual); Study Completion 2021-10-31 (Actual)

PRIMARY OUTCOMES:
muscle stiffness | baseline
  the examiners assess the mechanical properties of the fascial and soft tissues with a myoton
muscle stiffness | After treatment immediately "1 hour"
  the examiners assess the mechanical properties of the fascial and soft tissues with a myoton
muscle stiffness | After treatment, one week follow-up
  the examiners assess the mechanical properties of the fascial and soft tissues with a myoton

SECONDARY OUTCOMES:
Pain intensity | Baseline
  the examiners assess the pain intensity using a visual analoigue scale
Pain intensity | After treatment immediately "1 hour"
  the examiners assess the pain intensity using a visual analoigue scale
Pain intensity | After treatment, "one week follow-up"
  the examiners assess the pain intensity using a visual analoigue scale
Range of motion | Baseline
  the examiners assess the shoulder range of motion with an universal goniometer
Range of motion | After treatment immediately "1 hour"
  the examiners assess the shoulder range of motion with an universal goniometer
Range of motion | After treatment, "one week follow-up"
  the examiners assess the shoulder range of motion with an universal goniometer
Extensibility | Baseline
  the examiners assess the extensibility of the posterior part of the tissues of the shoulder using a digital inclinometer
Extensibility | After treatment immediately "1 hour"
  the examiners assess the extensibility of the posterior part of the tissues of the shoulder using a digital inclinometer
Extensibility | After treatment, "one week follow-up"
  the examiners assess the extensibility of the posterior part of the tissues of the shoulder using a digital inclinometer

CONTACTS AND LOCATIONS:
Overall Officials: Luis Ceballos Laita, PhD, Study Director — University of Valladolid
Locations (1):
- Sandra Jiménez Jiménez-del-Barrio, Soria, Spain

IPD SHARING:
Plan to Share IPD: No